CLINICAL TRIAL: NCT06301009
Title: The AI-CAC Model for Subclinical Atherosclerosis Detection on Chest X-ray: Prospective Validation Study (AI-CAC-PVS)
Brief Title: The AI-CAC Model for Subclinical Atherosclerosis Detection on Chest X-ray
Acronym: AI-CAC-PVS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Compagnia di San Paolo (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, MD, PhD, A.O.U. Città della Salute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AI-CAC-PVS
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Artery Calcification
Keywords: coronary artery calcium; chest x-ray; atherosclerotic cardiovascular disease; primary prevention; risk prediction; artificial intelligence
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-CAC arm (Experimental): All patients included in the study and undergoing AI-CAC calculation on a chest x-ray
  Interventions: Diagnostic Test: AI-CAC score

INTERVENTIONS:
Diagnostic Test: AI-CAC score — Deep-learning based prediction of the coronary artery calcium score with a plain chest x-ray

SUMMARY:
The AI-CAC model is an artificial intelligence system capable of assessing the presence of subclinical atherosclerosis on a simple chest radiograph. The present study will provide prospective validation of its diagnostic performance in a primary prevention population with a clinical indication for coronary artery calcium (CAC) testing.

DETAILED DESCRIPTION:
The AI-CAC-PVS project is a prospective, multicenter, single-arm clinical study, with enrollment at 5 Radiology Units in Piedmont (Italy). Consecutive individuals without prior reported cardiovascular events referred for a non-contrast chest CT for the assessment of coronary artery calcium (CAC) score for cardiovascular risk stratification purposes will be considered for inclusion in the study. Individuals who agree to participate in the study will undergo a standard chest radiograph, as the only deviation from clinical practice. The CAC score will be calculated on chest CT scans according to international standards, and the result will be provided to the patient. Any subsequent changes in behavioral habits, lipid-lowering, antiplatelet, antihypertensive, and antidiabetic therapies prescribed by the attending physician will be collected in a dedicated dataset, along with the occurrence of cardiovascular events at the last available follow-up.

The AI-CAC model will be applied to the chest radiograph, yielding an AI-CAC value as output. The patient, radiologist, and attending physician will not be informed of the AI-CAC value until the end of the study.

The primary outcome will be the accuracy of the AI-CAC model to detect the presence of subclinical atherosclerosis on chest x-ray as compared to the CT scan (i.e. CAC >0). The ability to predict clinical outcomes at follow-up (ASCVD, atherosclerotic cardiovascular disease events comprising myocardial infarction, ischemic stroke, coronary revascularization and cardiovascular death) will be assessed as exploratory secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Age between 40 and 75 years
* Clinical indication from the treating physician to undergo chest CT for CAC score evaluation

Exclusion Criteria:

* Prior cardiovascular events (myocardial infarction, coronary revascularization, transient ischemic attack, stroke, symptomatic peripheral vascular disease, arterial revascularization of peripheral districts)
* Cancer or other chronic diseases with an estimated prognosis of less than five years
* Technical contraindications to the execution of chest CT with electrocardiographic gating (highly penetrant atrial fibrillation, frequent ventricular extrasystoles)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the AI-CAC score to identify the presence of subclinical atherosclerosis on chest x-ray | Through study completion (anticipated average follow-up of 1 year).
  Diagnostic accuracy of the AI-CAC score to identify the presence of subclinical atherosclerosis (i.e. AI-CAC >0) on chest x-ray as compared to CAC measured on a non-contrast ECG-gated CT scan (i.e. CAC >0).
  The area under the curve (AUC) method will be used to evaluate the primary outcome.

SECONDARY OUTCOMES:
Percentage of individuals with a therapeutic management change by the attending physician based on the CAC score, with concordant AI-CAC. | Through study completion (anticipated average follow-up of 1 year).
  Potential impact on the implementation of primary prevention strategies: i.e. percentage of individuals with a therapeutic management change by the attending physician (increase or decrease in lipid-lowering therapy, initiation or discontinuation of antiplatelet therapy, behavioral measures) based on the CAC score, with concordant AI-CAC.
Comparison of ASCVD events occurring in patients without (AI-CAC=0) vs. with subclinical atherosclerosis (AI-CAC >0) based on the AI-CAC score, as assessed by Kaplan Meier estimates of ASCVD events occurring until study completion. | Through study completion (anticipated average follow-up of 1 year).
  Predictive ability of the AI-CAC score for the incidence of adverse cardiovascular events (myocardial infarction, stroke, cardiovascular death, or coronary revascularization) at the last available follow-up.

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed cardiovascular journal